CLINICAL TRIAL: NCT07314814
Title: Genetic Hallmarks of Patients With Congenital Portosystemic Shunts and Portopulmonary Hypertension
Acronym: Gen-PoPH-CPSS
Status: Not yet recruiting | Type: Observational
Sponsor: Prof. Valérie Mc Lin (Other)
Responsible Party: Sponsor-Investigator, Prof. Valérie Mc Lin, Prof. Dr. Med., University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Other Study IDs: 2024-01698; 2024-01698 (Other: Commission Cantonale d'Ethique de la Recherche (CCER) , Geneva Switzerland)
Record Dates: First submitted 2025-12-18; First posted 2026-01-02 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Portopulmonary Hypertension; Pulmonary Arterial Hypertension (PAH); Congenital Portosystemic Shunt
Keywords: CPSS; PoPH; PAH; Genetic; Genomic; IRCPSS
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Congenital Portosystemic Shunt | interventions — Genome-Wide Association Study

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood sample -> genomic DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 30 families: patient + parents+ siblings
  Interventions: Genetic: targeted gene panels analysis; Genetic: whole genome analysis

INTERVENTIONS:
Genetic: targeted gene panels analysis — The following gene panels will be analyzed : pulmonary arterial hypertension ; hereditary hemorrhagic telangiectasia ; congenital heart disease and potentially pathogenic variants in genes previously associated with PoPH in cirrhosis cohort.
Genetic: whole genome analysis — Family-based identification of dominant or recessive potentially pathogenic variants.

SUMMARY:
Congenital portosystemic shunt (CPSS) are rare vascular malformations causing blood from the intestines to bypass the liver and directly flow into body's general circulation. Such liver bypass can cause several health problems, one of the most severe being portopulmonary hypertension (PoPH).

The goal of this study is to identify pathogenic and potentially pathogenic genetic variants in patients who have both CPSS and PoPH. Future research will assess the contribution of these genetic variants to the development of PoPH.

The long-term goal is to use genetic information to identify patients with congenital portosystemic shunts (CPSS) or chronic liver disease who are at risk of developing PoPH to offer anticipatory management.

Children and adult patients with both CPSS and PoPH, as well as their close relatives (patient's parents and siblings) can take part in the study. Genetic variations within each family will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a participant to the IRCPSS with history of PoPH
* Trios composed of CPSS PoPH patients and their parents (trios are mandatory)
* Brother/sister of an enrolled patient
* Trios accept to provide biological samples (blood), sign the inform consent.
* Siblings and/or siblings' legal representatives accept to provide biological samples (blood), sign the inform consent.

Exclusion Criteria:

* Trio condition is not met.
* No genuine parent-offspring trios (check for medically assisted procreation with donors, and adoption)
* For siblings, half-brothers or half-sisters are excluded, as well as adopted children, or children issued from medically assisted procreation with donors.
* Secondary portosystemic shunts
* The refusal by the patient or the patient's legal representatives to provide biological samples or agree with the proposed procedure or after voluntary withdrawal from the project.
* The refusal of one of the parents to provide biological samples or to agree with the proposed procedure or after voluntary withdrawal from the project.

Ages: 1 Day to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patient participant in the IRCPSS, with history of CPSS and PoPH ; both parents of the patient participants; possibly patient siblings.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
List of variants from targeted analysis of selected gene panels | From February 2026 to February 2029
  presence/absence of pathogenic variants in known genes (pulmonary arterial hypertension ; hereditary hemorrhagic telangiectasia ; congenital heart disease) and potentially pathogenic variants in genes previously associated with PoPH in cirrhosis cohort.
List of variants from whole genome analysis | Fron February 2026 to August 2029
  variants identified using family based search for dominant or recessive potentially pathogenic variants

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Geneva / University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
to be determined